CLINICAL TRIAL: NCT05813925
Title: Efficacy and Safety of Cagrilintide S.C. 2.4 mg in Combination With Semaglutide S.C. 2.4 mg (CagriSema S.C. 2.4 mg/2.4 mg) Once-Weekly in East Asian Participants With Overweight or Obesity
Brief Title: A Research Study to See How Well CagriSema Helps People in East Asia With Excess Body Weight Lose Weight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4762; U1111-1277-3764 (Other: World Health Organization (WHO)); jRCT2031220734 (Registry Identifier: jRCT (Japan))
Record Dates: First submitted 2023-04-03; First posted 2023-04-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Obesity or Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- CagriSema 2.4 mg/2.4 mg (Experimental): Participants will receive 2.4 milligrams (mg) cagrilintide and 2.4 mg semaglutide subcutaneously (s.c.) once-weekly (OW) after a dose escalation period of 16 weeks (0.25 mg of cagrilintide and 0.25 mg of semaglutide from weeks 0-4, 0.5 mg of cagrilintide and 0.5 mg of semaglutide from weeks 5-8, 1 mg of cagrilintide and 1 mg of semaglutide from weeks 9-12 and 1.7 mg of cagrilintide and 1.7 mg of semaglutide from weeks 13-16) during the maintenance period for 52 weeks
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Semaglutide 2.4 mg (Active Comparator): Participants will receive semaglutide s.c. 2.4 mg and placebo matched to semaglutide OW after a dose escalation period of 16 weeks (0.25 mg for weeks 0-4, 0.5 mg for weeks 5-8, 1 mg for weeks 9-12 and 1.7 mg for weeks 13-16) during the maintenance period for 52 weeks
  Interventions: Drug: Semaglutide; Drug: Placebo Semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive 2.4 mg cagrilintide s.c. OW after a dose escalation period of 16 weeks for 52 weeks
  Arms: CagriSema 2.4 mg/2.4 mg
Drug: Semaglutide — Participants will receive 2.4 mg semaglutide s.c. OW after a dose escalation period of 16 weeks for 52 weeks
Drug: Placebo Semaglutide — Participants will receive placebo matched to semaglutide
  Arms: Semaglutide 2.4 mg

SUMMARY:
This study will look at how well the new medicine CagriSema helps people with excess body weight lose weight compared to another medicine, semaglutide. The participants will receive one injection once a week. The study medicine will be injected with a thin needle, typically in the stomach, thighs or upper arms. The study will last for about 1½ years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age greater than to or equal 18 years at the time of signing informed consent
* a) Body mass index (BMI) greater than or equal to 27.0 kilograms per square meter (kg/m^2) with greater than or equal to 2 obesity-related complications or b) BMI greater than or equal to 35.0 kg/m^2 with greater than or equal to 1 obesity-related complication. At least one complication should be hypertension, dyslipidaemia or T2D

Diabetes-related for participant with T2D

* Diagnosed with T2D greater than or equal to 180 days before screening
* HbA1c 7.0-10.0 percent (53-86 millimoles per mole [mmol/mol]) (both inclusive) as measured by central laboratory at screening
* Treatment with either lifestyle intervention, or treatment with 1-3 marketed oral antidiabetic drugs (OAD)s (metformin, α-glucosidase inhibitors [AGI], glinides, sodium-glucose cotransporter 2 inhibitor [SGLT2i]), thiazolidinediones, or sulphonylureas [SU] as a single agent or in combination) according to local label
* Treatment with oral antidiabetic drugs should be stable (same drug(s), dose and dosing frequency) for at least 90 days before screening

Exclusion Criteria:

Obesity-related

- Treatment with any medication prescribed for the indication of obesity or weight management within 90 days before screening

Glycaemia-related for participant without T2D

* HbA1c greater than or equal to 6.5 percent (48 mmol/mol) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes

Diabetes-related for participant with T2D

* Renal impairment with estimated glomerular filtration rate (eGFR) lesser than 30 milli liter per min/1.73 meter square (mL/min/1.73 m^2) as measured by central laboratory at screening
* Clinically significant or severe hypoglycaemia within 6 months of screening or history of hypoglycaemia unawareness
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by a fundus examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Relative Change in Body Weight | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)

SECONDARY OUTCOMES:
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 20 Percent | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants
Change in Waist Circumference Measured According to Japan Society for the Study of Obesity (JASSO) Guideline | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeter (cm)
Change in Visceral Fat Area (VFA) Measured by CT Scan in Subset of the Japanese Study Population | From baseline (week 0) to end of treatment (week 68)
  Measured as percentage point
Change in VFA Measured by CT Scan in Subset of the Japanese Study Population | From baseline (week 0) to end of treatment (week 68)
  Measured in centimeter square (cm^2)
Number of Participants Who Achieve (Yes/No): VFA lesser than 100 cm^2 (Only for Participants with VFA greater than or equal to 100 cm^2 at Baseline) | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 25 Percent | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 15 Percent | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants
Number of Participants Who Achieve (Yes/No): Body Weight Reduction Greater Than or Equal to 10 Percent | From baseline (week 0) to end of treatment (week 68)
  Measured as count of participants
Relative Change in Body Weight | From baseline (week 0) to week 20
  Measured in percentage (%)
Change in Body Weight | From baseline (week 0) to end of treatment (week 68)
  Measured in kilogram (kg)
Change in Body Mass Index (BMI) | From baseline (week 0) to end of treatment (week 68)
  Measured in kilogram per meter square (kg/m^2)
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage points
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 68)
  Measured as millimole per liter (mmol/L)
Change in Fasting Insulin | From baseline (week 0) to end of treatment (week 68)
  Measured as milliunits per liter (mU/L)
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeter of mercury (mmHg)
Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 68)
  Measured in millimeter of mercury (mmHg)
Change in Total Cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
Change in High-Density Lipoprotein (HDL) Cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
Change in Low-Density Lipoprotein (LDL) Cholesterol | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
Change in Very Low-Density Lipoprotein (VLDL) | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
Change in Triglycerides | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
Change in Free fatty Acids | From baseline (week 0) to end of treatment (week 68)
  Measured in percentage (%)
Change in Impact of Weight on Quality of Life-Lite for clinical trials (IWQOL-Lite-CT) Physical Function Score | From baseline (week 0) to end of treatment (week 68)
  IWQOL-Lite-CT is a 20-item patient reported outcome (PRO) instrument used to assess the impact of body weight changes in obesity studies on patient's physical and psychosocial functioning in three composite scores (physical function, physical and psychosocial) and a total score
Number of Treatment-Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of study (week 75)
  Measured as count of events
Number of Serious Adverse Events (SAEs) | From baseline (week 0) to end of study (week 75)
  Measured as count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency' (dept. 2834), Study Director — Novo Nordisk A/S
Locations (28):
- Japan (27):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Fukushima, Japan
  - Tsuruma Kaneshiro Diabetes Clinic_Internal medicine, Yamato-shi, Kanagawa
  - Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - OCROM Clinic_Internal medicine, Suita-shi, Osaka
  - Yao Tokushukai General Hospital_Cardiovascular division, Yao-shi, Osaka
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - The University of Tokyo Hospital, Diabetes and Metabolic, Bunkyo-ku, Tokyo
  - Akaicho Clinic, Chiba-shi, Chiba
  - Suidoubashi Medical Clinic_Internal Medicine, Chiyoda-ku, Tokyo
  - The Institute of Medical Science, Asahi Life Foundation_Internal Medicine, Chuo-ku, Tokyo
  - The Institute of Medical Science, Asahi Life Foundation, Chuo-ku, Tokyo
  - Okabe Clinic, Chuo-ku, Tokyo
  - Kawada Clinic, Gunma
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Naka Kinen Clinic, Ibaraki
  - Iwate Medical University Uchimaru Medical Center, Division of Diabetes and Metabolism and Endocrine medicine, Numakunai
  - Osaka NISHI-UMEDA Clinic_Internal Medicine, Osaka
  - Osaka NISHI-UMEDA Clinic, Osaka
  - Shinsapporo Seiryou Hospital, General Clinical Department, Sapporo-shi, Hokkaido
  - Shinden Higashi Clinic_Internal medicine, Sendai-shi, Miyagi
  - Shinden Higashi Clinic, Sendai-shi, Miyagi
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
  - ToCROM Clinic_Internal Medicine, Tokyo
  - Minamino Cardiovascular Hospital_Cardiovascular medicine, Tokyo
- National Taiwan University Hospital_main, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com